CLINICAL TRIAL: NCT03331198
Title: An Open-Label, Phase 1/2 Study of JCAR017 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma (017004)
Brief Title: Study Evaluating Safety and Efficacy of JCAR017 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juno Therapeutics, a Subsidiary of Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017004; TRANSCEND-CLL-004 (Other: Juno Therapeutics, Inc.)
Record Dates: First submitted 2017-10-29; First posted 2017-11-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Small Lymphocytic
Keywords: TRANSCEND_CLL_004
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Intervention Model Description: Phase 1: subjects will be assigned to receive JCAR017, or JCAR017 + ibrutinib, or JCAR017 + venetoclax Phase 2: subjects will be assigned to receive JCAR017 at the recommended dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 JCAR017 monotherapy (Experimental): Subjects will be assigned to receive JCAR017 (lisocabtagene maraleucel)
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel)
- Phase 1 JCAR017 + ibrutinib (Experimental): Subjects receiving ibrutinib at baseline will be assigned to receive JCAR017 (lisocabtagene maraleucel) at the recommended dose from the Phase 1 monotherapy arm + ibrutinib
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel) + ibrutinib
- Phase 2 JCAR017 monotherapy (Experimental): Subjects will receive JCAR017 (lisocabtagene maraleucel) at the recommended dose from the Phase 1 monotherapy arm
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel)
- Phase 1 JCAR017 + venetoclax (Experimental): Subjects will receive venetoclax as bridging anticancer therapy until lymphodepletion chemotherapy/ JCAR017 (lisocabtagene maraleucel) at the recommended dose from the Phase 1 monotherapy arm. After JCAR017 infusion subjects will receive venetoclax until Day 90.
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel) + venetoclax
- Phase 2 JCAR017 Double-Exposed Monotherapy Expansion (DEME) (Experimental): Subjects will receive JCAR017 monotherapy
  Interventions: Biological: JCAR017 (lisocabtagene maraleucel)

INTERVENTIONS:
Biological: JCAR017 (lisocabtagene maraleucel) — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCAR017. During JCAR017 production, participants may receive bridging anticancer therapy for disease control. Treatment will include lymphodepleting chemotherapy followed by one dose of JCAR017 administered by intravenous (IV) injection.
  Arms: Phase 1 JCAR017 monotherapy; Phase 2 JCAR017 Double-Exposed Monotherapy Expansion (DEME); Phase 2 JCAR017 monotherapy
Biological: JCAR017 (lisocabtagene maraleucel) + ibrutinib — Participants eligible for this cohort should be receiving ibrutinib at the time of screening. For participants who previously discontinued ibrutinib, ibrutinib will be started as soon as possible after eligibility is confirmed. Ibrutinib treatment will continue for up to 90 days after JCAR017 infusion (or longer for participants who are receiving benefit from ibrutinib). Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCAR017. During JCAR017 production, participants may receive bridging chemotherapy for disease control. Upon successful generation of JCAR017 product, participants will receive treatment with JCAR017 therapy. Each cycle will include lymphodepleting chemotherapy followed by one dose of JCAR017 administered by intravenous (IV) injection.
  Arms: Phase 1 JCAR017 + ibrutinib
Biological: JCAR017 (lisocabtagene maraleucel) + venetoclax — Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of JCAR017. During JCAR017 production, participants will receive venetoclax as bridging anticancer therapy on a weekly ramp up dosing schedule until stopping one day prior to lymphodepletion. Treatment will include lymphodepleting chemotherapy followed by one dose of JCAR017 administered by intravenous (IV) injection, and the day after infusion venetoclax will be re-initiated.
  Arms: Phase 1 JCAR017 + venetoclax

SUMMARY:
This is a Phase 1/2, open-label, multicenter study to determine the efficacy and safety of JCAR017 in adult subjects with relapsed or refractory CLL or SLL. The study will include a Phase 1 part to determine the recommended dose of JCAR017 monotherapy in subjects with relapsed or refractory CLL or SLL, followed by a Phase 2 part to further assess the efficacy and safety of JCAR017 monotherapy treatment at the recommended dose. A separate Phase 1 cohort will assess the combination of JCAR017 and concurrent ibrutinib. Another separate Phase 1 cohort will assess the combination of JCAR017 and concurrent venetoclax. In all subjects, the safety, efficacy, and pharmacokinetics (PK) of JCAR017 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of:

  1. CLL with an indication for treatment based on the Investigator's opinion and measurable disease, or
  2. SLL (lymphadenopathy and/or splenomegaly and < 5×10^9 CD19+ CD5+ clonal B lymphocytes/L [< 5000/µL] in the peripheral blood at diagnosis with measurable disease that is biopsy-proven SLL)
* Subjects (other than those in the ibrutinib + JCAR017 combination therapy and DEME cohort) must have received and failed Bruton tyrosine kinase inhibitor (BTKi) treatment or have been deemed ineligible for BTKi therapy.
* Subjects in the JCAR017 monotherapy cohorts must have received previous treatment as follows:

  1. Monotherapy cohorts EXCEPT DEME cohort: Subjects with CLL or SLL and high-risk features must have failed at least 2 lines of prior therapy.
  2. Monotherapy cohorts EXCEPT DEME cohort: Subjects with CLL or SLL and standard-risk features must have failed at least 3 lines of prior therapy.
  3. DEME cohort ONLY: Subjects with relapsed or refractory CLL or SLL, irrespective of cytogenetic risk features, must have received at least 2 lines of prior therapy including a BTKi and a BCL2i.
* Subjects in the ibrutinib + JCAR017 combination therapy cohort must either:

  1. be receiving ibrutinib and progressing at the time of study enrollment
  2. be receiving ibrutinib for at least 6 months with a response less than complete response/remission (CR) and have high-risk features as defined in inclusion criterion 5a
  3. have BTK or PLCgamma2 mutations per local laboratory assessment, with or without progression on ibrutinib
  4. have previously received ibrutinib and have no contraindications to restarting ibrutinib
* Eastern Cooperative Oncology Group performance status of ≤ 1
* Assessed by the Investigator to have adequate bone marrow function to receive lymphodepleting chemotherapy
* Adequate organ function, defined as:

  1. Serum creatinine ≤ 1.5 × age-adjusted upper limit of normal (ULN) OR calculated creatinine clearance > 30 mL/min
  2. Alanine aminotransferase ≤ 5 × ULN and total bilirubin < 2.0 mg/dL (or < 3.0 mg/dL for subjects with Gilbert's syndrome or leukemic infiltration of the liver)
  3. Adequate pulmonary function, defined as ≤ Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 dyspnea and saturated oxygen (SaO2) ≥ 92% on room air
  4. Adequate cardiac function, defined as left ventricular ejection fraction ≥ 40% as assessed by echocardiogram or multiple uptake gated acquisition scan performed within 30 days prior to determination of eligibility
* Subject either currently has central vascular access or is a candidate to receive central vascular access or peripheral vascular access for leukapheresis procedure.
* If prior CD19-targeted therapy has been administered, subject must have CD19-positive disease confirmed by immunohistochemistry or flow cytometry since completing the prior CD19-targeted therapy.
* Subjects in ibrutinib + JCAR017 combination cohort must have progressed on a BTKi and have received prior therapy with venetoclax
* Subjects in venetoclax + JCAR017 combination cohort must:

  1. have failed at least 1 prior line of therapy, including failed BTKi therapy or have been deemed ineligible to receive BTKi
  2. be venetoclax naive (required for dose expansion) or
  3. if prior venetoclax (only for dose escalation)
  4. have no contraindictions to re-initiation of venetoclax based on prior intolerance and have had at least 6 months elapsed since the last dose of venetoclax, if either, best response was stable disease, or subject experienced disease progression on venetoclax, or within 6 months of venetoclax discontinuation
* subjects in the venetoclax + JCAR017 combination must have hemoglobin >=9 g/dL, absolute neutrophil count >=500mm3 and platelets>= 75,000/mm3, unless cytopenias are judged by investigator to be due to CLL infiltration of the bone marrow
* must have diagnosis of CLL or SLL with an indication for treatment based on the investigator's opinion and measurable disease (any of the following measurable lymph nodes ≥1.5 cm in the greatest transverse diameter and/or hepatomegaly or splenomegaly) and demonstration of CLL cells in the peripheral blood by flow cytometry

Exclusion Criteria:

* Subjects with known active central nervous system (CNS) involvement by malignancy. Those with prior CNS disease that has been effectively treated will be eligible if treatment was completed at least 3 months prior to enrollment with no evidence of symptomatic disease and stable abnormalities on repeat imaging.
* History of another primary malignancy that has not been in remission for at least 2 years. (The following are exempt from the 2-year limit: nonmelanoma skin cancer, completely resected stage 1 solid tumor with low risk for recurrence, curatively treated localized prostate cancer, cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Pap smear, and in situ breast cancer that has been completely resected.)
* Subjects with Richter's transformation
* Prior treatment with any gene therapy product
* Active hepatitis B, active hepatitis C, or active human immunodeficiency virus (HIV) infection
* Systemic fungal, bacterial, viral, or other infection that is not controlled
* Presence of acute or extensive chronic graft versus host disease (GVHD)
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
* History or presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, aphasia, stroke with current neurologic sequelae, severe brain injuries, dementia, Parkinson's disease, cerebellar disease,cerebral edema, or psychosis
* Pregnant or nursing (lactating) women
* Use of any of the following medications or treatments within the noted time prior to leukapheresis:

  1. Alemtuzumab within 6 months prior to leukapheresis
  2. Allogeneic hematopoietic stem cell transplant within 100 days prior to leukapheresis
  3. Cladribine within 3 months prior to leukapheresis
  4. Donor lymphocyte infusions (DLI) within 2 months prior to leukapheresis
  5. Radiation including large bone marrow fields such as sternum or pelvis within 6 weeks prior to leukapheresis
  6. Fludarabine within 4 weeks prior to leukapheresis
  7. GVHD therapies such as calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate mofetil, rapamycin, or immunosuppressive antibodies (such as anti-tumor necrosis factor-α [TNFα], anti-interleukin-6 [IL-6], or anti-interleukin-6 receptor [IL 6R]) within 4 weeks prior to leukapheresis
  8. Cyclophosphamide, ifosfamide, bendamustine, chlorambucil, or melphalan within 2 weeks prior to leukapheresis
  9. Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) within 7 days prior to leukapheresis
  10. Anti-CD20 monoclonal antibodies within 7 days prior to leukapheresis
  11. Venetoclax within 4 days prior to leukapheresis
  12. Idelalisib or duvelisib within 2 days prior to leukapheresis
  13. Lenalidomide or covalent and non-covalent BTKi within 1 day prior to leukapheresis
  14. Experimental agents, including off-label use of approved drugs (with the exception of acalabrutinib which may be continued up to the day before leukapheresis), within 4 weeks prior to leukapheresis unless progression is documented on the experimental therapy and at least 3 half-lives have elapsed prior to leukapheresis
* Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the Investigator; or subject unwillingness or inability to follow the procedures required in the protocol
* Progressive vascular tumor invasion, thrombosis, or embolism
* Deep vein thrombosis or embolism not managed on a stable regimen of anticoagulation
* Use of any of the following medications or treatments within the noted time prior to leukapheresis lenalidomide or acalabrutinib within 1 day prior to leukapheresis experimental agents, including off-label use of approved drugs, within 4 weeks prior to leukapheresis.
* Venous thrombosis or embolism requiring treatment but not managed on a stable regimen of anticoagulation
* For subjects in the venetoclax + JCAR017 combination cohorts only, concomitant treatment with CYP3A moderate/strong inducers or moderate/strong inhibitors which cannot be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2027-11-26 (Estimated); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Phase 1 JCAR017 monotherapy arm: adverse events | Up to 48 months post treatment
  Proportion of subjects experiencing adverse events
Phase 1 JCAR017 monotherapy arm: laboratory abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 1 JCAR017 and ibrutinib combination dose escalation therapy arm: adverse events | Up to 48 months post treatment
  Proportion of subjects experiencing adverse events
Phase 1 JCAR017 and ibrutinib combination dose escalation therapy arm: laboratory abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm | Through post treatment up to Month 48
  Proportion of subjects who have CR after treatment with JCAR017 + ibrutinib using iwCLL 2018 guidelines
Phase 1 JCAR017 and venetoclax combination dose escalation therapy arm: adverse events | Up to 48 months post treatment
  Proportion of subjects experiencing adverse events
Phase 1 JCAR017 and venetoclax combination dose escalation therapy arm: laboratory abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm | Through post treatment up to Month 48
  Proportion of subjects who have CR after treatment with JCAR017 + venetoclax using iwCLL 2018 guidelines
Phase 2 JCAR017 monotherapy expansion arm | Through post treatment up to Month 48
  Proportion of subjects who have CR after treatment with JCAR017 using iwCLL 2018 guidelines
Phase 2 JCAR017 Double exposed monotherapy expansion arm: overall response rate (ORR) | Up to approximately 24 months
  ORR defined as the rate of complete response/remission (CR) [including complete response/remission with incomplete marrow recovery (Cri)] plus PR [including nodular partial response (nPR)] based on Independent Review Committee (IRC) assessment using International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines

SECONDARY OUTCOMES:
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: adverse events | Up to 48 months post treatment
  Proportion of subjects experiencing adverse events
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: laboratory abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: ORR | Up to 48 months post treatment
  Defined as the rate of CR (including CRi)
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: MRD negative response rate in peripheral blood | Up to 48 months post treatment
  Proportion of subjects who achieve MRD CR
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: MRD-negative CR rate in peripheral blood | Up to 48 months post treatment
  Proportion of subjects who achieve MRD CR
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: Duration of response (DOR) | Up to 48 months post treatment
  Defined as the time from first response (CR, CRi, nPR, or PR) to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: Duration of complete response (DoCR) | Up to 48 months post treatment
  Defined as the time from first CR or CRi to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: Time to response (TTR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR, CRi, nPR, or PR
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: Time to complete response (TTCR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: PFS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and ibrutinib combination dose expansion therapy arm: OS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the date of death due to any cause
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: adverse events | Up to 48 months post treatment
  Proportion of subject experiencing adverse events
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: lab abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: ORR | Through post treatment Day 90
  Defined as the rate of CR (including CRi)
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: MRD-negative response rate in peripheral blood | Up to 48 months post treatment
  Proportion of subjects who achieve MRD CR
Phase 1 JCAR017 and venetoclax combination dose escalation therapy arm: MRD-negative CR rate in peripheral blood | Through post treatment Day 90
  Proportion of subjects who achieve MRD CR
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: Duration of response (DOR) | Up to 48 months post treatment
  Defined as the time from first response (CR, CRi, nPR, or PR) to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: Duration of complete response (DoCR) | Up to 48 months post treatment
  Defined as the time from first CR or CRi to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: Time to response (TTR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR, CRi, nPR, or PR
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: Time to complete response (TTCR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: PFS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the earlier date of PD or death due to any cause
Phase 1 JCAR017 and venetoclax combination dose expansion therapy arm: OS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the date of death due to any cause
Phase 2 JCAR017 Monotherapy Expansion Arm: adverse events | Up to 48 months post treatment
  Proportion of subjects experiencing adverse events
Phase 2 JCAR017 Monotherapy Expansion Arm: laboratory abnormalities | Up to 48 months post treatment
  Proportion of subjects experiencing laboratory abnormalities
Phase 2 JCAR017 Monotherapy Expansion Arm: ORR | Up to 48 months post treatment
  Defined as the rate of CR (including CRi)
Phase 2 JCAR017 Monotherapy Expansion Arm: MRD negative response rate in peripheral blood | Up to 48 months post treatment
  Proportion of subjects who achieve MRD CR
Phase 2 JCAR017 Monotherapy Expansion Arm: MRD-negative CR rate in peripheral blood | Up to 48 months post treatment
  Proportion of subjects who achieve MRD CR
Phase 2 JCAR017 Monotherapy Expansion Arm: Duration of response (DOR) | Up to 48 months post treatment
  Defined as the time from first response (CR, CRi, nPR, or PR) to the earlier date of PD or death due to any cause
Phase 2 JCAR017 Monotherapy Expansion Arm: Duration of complete response (DoCR) | Up to 48 months post treatment
  Defined as the time from first CR or CRi to the earlier date of PD or death due to any cause
Phase 2 JCAR017 Monotherapy Expansion Arm: Time to response (TTR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR, CRi, nPR, or PR
Phase 2 JCAR017 Monotherapy Expansion Arm: Time to complete response (TTCR) | Up to 48 months post treatment
  Defined as the interval from JCAR017 infusion to the first documentation of CR
Phase 2 JCAR017 Monotherapy Expansion Arm: PFS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the earlier date of PD or death due to any cause
Phase 2 JCAR017 Monotherapy Expansion Arm: OS | Up to 48 months post treatment
  Defined as the time from JCAR017 infusion to the date of death due to any cause
Phase 2 JCAR017 Monotherapy Expansion Arm: Health-related quality of life (HRQoL) questionnaire | Up to 48 months post treatment
  Change from baseline in HRQoL assessed using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30
Phase 2 JCAR017 Monotherapy Expansion Arm: HRQoL questionnaire | Up to 48 months post treatment
  Change from baseline in HRQoL assessed using the EORTC chronic lymphocytic leukemia (CLL)-specific module QLQ-CLL-17
Phase 2 JCAR017 Monotherapy Expansion Arm: Health economics and outcomes research (HEOR) questionnaire | Up to 48 months post treatment
  Change from baseline in measurement of health utility values using EuroQol instrument EQ-5D-5L
Phase 2 JCAR017 Monotherapy Expansion Arm: HEOR questionnaire | Up to 48 months post treatment
  Proportion of participants with intensive care unit (ICU) inpatient days
Phase 2 JCAR017 Monotherapy Expansion Arm: HEOR questionnaire | Up to 48 months post treatment
  Proportion of participants with non-ICU inpatient days
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: adverse events | Up to approximately 24 months
  Proportion of subjects experiencing adverse events
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: laboratory abnormalities | Up to approximately 24 months
  Proportion of subjects experiencing laboratory abnormalities
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: Duration of response (DOR) | Up to approximately 24 months
  Defined as the time from first response (CR, CRi, nPR, or PR) to the earlier date of PD or death due to any cause
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: CR rate | Up to approximately 24 months
  Defined as the rate of CR (including CRi) based on IRC assessment using iwCLL 2018 guidelines
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: MRD-negative response rate in peripheral blood | Up to approximately 24 months
  Proportion of subjects who achieve MRD negative status
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: MRD-negative CR rate in peripheral blood | Up to approximately 24 months
  Proportion of subjects who achieve MRD-negative CR
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: Time to response (TTR) | Up to approximately 24 months
  Defined as the interval from JCAR017 infusion to the first documentation of CR, CRi, nPR, or PR
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: Time to complete response (TTCR) | Up to approximately 24 months
  Define as the interval from JCAR017 infusion to the first documentation of CR
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: Progression free survival (PFS) | Up to approximately 24 months
  Defined as the time from JCAR017 infusion to the earlier date of PD or death due to any cause
Phase 2 JCAR017 Double-Exposed Monotherapy Expansion Arm: Overall Survival (OS) | Up to approximately 24 months
  Defined as the time from JCAR017 infusion to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (83):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - City Of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University Of California San Diego Moores Cancer Center, La Jolla, California
  - Local Institution - 0059, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Local Institution - 0010, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Local Institution - 0110, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Local Institution - 0085, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Local Institution - 0104, Atlanta, Georgia
  - Local Institution - 0019, Atlanta, Georgia
  - The Blood and Marrow Transplant Group of Georgia (BMTGA), Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University Of Chicago Medical Center, Chicago, Illinois
  - Franciscan St. Francis Health - Indiana Blood and Marrow Transplantation (IBMT), Indianapolis, Indiana
  - Local Institution - 0107, Wichita, Kansas
  - Norton Healthcare - Norton Cancer Institute, Louisville, Kentucky
  - Local Institution - 0027, New Orleans, Louisiana
  - Local Institution - 0005, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Local Institution - 0015, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University Of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Local Institution - 0062, Detroit, Michigan
  - Local Institution - 0109, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - Basking Ridge, Basking Ridge, New Jersey
  - Astera Cancer Care, Edison, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Local Institution - 0077, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Local Institution - 0035, New York, New York
  - Columbia University Medical Center, New York, New York
  - Local Institution - 0026, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Seidman Cancer Center (Case Western), Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center (Stephenson Cancer Center), Oklahoma City, Oklahoma
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Local Institution - 0098, Eugene, Oregon
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Local Institution - 0029, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Local Institution - 0083, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Local Institution - 0079, Dallas, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Local Institution - 0028, Salt Lake City, Utah
  - Local Institution - 0113, Charlottesville, Virginia
  - Local Institution - 0087, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Local Institution - 0018, Seattle, Washington
  - Froedtert Hospital BMT Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Local Institution - 0112, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- [Derived] Siddiqi T, Maloney DG, Kenderian SS, Brander DM, Dorritie K, Soumerai J, Riedell PA, Shah NN, Nath R, Fakhri B, Stephens DM, Ma S, Feldman T, Solomon SR, Schuster SJ, Perna SK, Tuazon SA, Ou SS, Papp E, Peiser L, Chen Y, Wierda WG. Lisocabtagene maraleucel in chronic lymphocytic leukaemia and small lymphocytic lymphoma (TRANSCEND CLL 004): a multicentre, open-label, single-arm, phase 1-2 study. Lancet. 2023 Aug 19;402(10402):641-654. doi: 10.1016/S0140-6736(23)01052-8. Epub 2023 Jun 6. PMID 37295445
- [Derived] Teoh J, Brown LF. Developing lisocabtagene maraleucel chimeric antigen receptor T-cell manufacturing for improved process, product quality and consistency across CD19+ hematologic indications. Cytotherapy. 2022 Sep;24(9):962-973. doi: 10.1016/j.jcyt.2022.03.013. Epub 2022 May 21. PMID 35610089
- [Derived] Siddiqi T, Soumerai JD, Dorritie KA, Stephens DM, Riedell PA, Arnason J, Kipps TJ, Gillenwater HH, Gong L, Yang L, Ogasawara K, Thorpe J, Wierda WG. Phase 1 TRANSCEND CLL 004 study of lisocabtagene maraleucel in patients with relapsed/refractory CLL or SLL. Blood. 2022 Mar 24;139(12):1794-1806. doi: 10.1182/blood.2021011895. PMID 34699592
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03331198.html